CLINICAL TRIAL: NCT04971395
Title: A Randomized, Double-blind, Placebo Controlled, First-in-Human Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of a Single Intravenous Infusion of XTMAB-16 in Healthy Adult Participants
Brief Title: Safety, Tolerability, and Pharmacokinetics of a Single Intravenous Infusion of XTMAB-16 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xentria, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: XTMAB-16-101
Record Dates: First submitted 2021-07-07; First posted 2021-07-21 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Single IV Infusion
  Interventions: Drug: Placebo
- XTMAB-16 2mg/kg (Experimental): Single IV Infusion
  Interventions: Drug: XTMAB-16 2 mg/kg
- XTMAB-16 4mg/kg (Experimental): Single IV Infusion
  Interventions: Drug: XTMAB-16 4mg/kg

INTERVENTIONS:
Drug: Placebo — Single dose of 2 or 4 mg/kg
  Arms: Placebo
Drug: XTMAB-16 2 mg/kg — Single dose of 2 mg/kg
  Arms: XTMAB-16 2mg/kg
Drug: XTMAB-16 4mg/kg — Single dose of 4 mg/kg
  Arms: XTMAB-16 4mg/kg

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled, first-in-human, single intravenous (IV) infusion of XTMAB-16 (formerly referred to as KBMAB-16) in normal healthy male and female participants.

DETAILED DESCRIPTION:
A total of 24 normal healthy adult participants will be enrolled and assigned into 2 treatment cohorts with 12 participants (9 on XTMAB-16 and 3 on placebo) in each cohort. Participants will receive a single IV infusion of 2 mg/kg or 4 mg/kg of XTMAB-16 or placebo on Day 1.

ELIGIBILITY:
Key Inclusion Criteria:

* The participant is a healthy adult male or female aged 18 to 45 years, inclusive, at the time of informed consent.
* The participant weighs between 45 kg (99 lbs) and 100 kg (220 lbs) and has a body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive, at the time of informed consent.
* The participant agrees to use highly effective method of contraception from the time of signing consent throughout 90 days after dosing.

Key Exclusion Criteria:

* The participant has received any investigational compound within 90 days before dosing.
* The participant has any clinically significant illness, such as cardiovascular, neurologic, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, endocrine, or psychiatric disease or disorder, or other abnormality, which may affect the participant's safety, increase risk of seizure or lower the seizure threshold, or potentially confound the study results. It is the responsibility of the Investigator to assess the clinical significance of any conditions the participant may have; however, consultation with the Xentria Medical Monitor may be warranted.
* The participant has a known hypersensitivity to any component of the formulation of XTMAB-16.
* The participant has a positive result for drugs of abuse (defined as any illicit drug use) or alcohol at Screening or Baseline (Day -2).
* The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to Screening or is unwilling to agree to abstain from alcohol and drugs throughout the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ray Goldwater, MDCM, M.Sc(A), CPI, Study Director — Parexel Baltimore Early Phase Clinical Unit
Locations (1):
- MedStar Harbor Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 24 normal healthy adult participants were planned to be enrolled and assigned into 2 treatment cohorts with 12 participants (9 on XTMAB-16 and 3 on placebo). Participants received a single IV infusion of 2 or 4 mg/kg of study drug (XTMAB-16 or placebo) on Day 1.
Groups:
- Pooled Placebo: Participants received a single IV Infusion of Placebo
- Single IV Infusion of 2 mg/kg of XTMAB-16: Participants received a single dose of 2 mg/kg of XTMAB-16
- Single IV Infusion of 4 mg/kg of XTMAB-16: Participants received a single dose of 4 mg/kg of XTMAB-16
Period: Overall Study
Arm/Group | Pooled Placebo | Single IV Infusion of 2 mg/kg of XTMAB-16 | Single IV Infusion of 4 mg/kg of XTMAB-16
Started | 6 | 10 | 9
Completed | 6 | 9 | 9
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Single IV Infusion of 2 mg/kg of XTMAB-16: Participants received a single dose of 2 mg/kg XTMAB-16
- Single IV Infusion of 4 mg/kg of XTMAB-16: Participants received a single dose of 4 mg/kg XTMAB-16
- Total: Total of all reporting groups
Arm/Group | Single IV Infusion of 2 mg/kg of XTMAB-16 | Single IV Infusion of 4 mg/kg of XTMAB-16 | Pooled Placebo | Total
Number analyzed (Participants) | 10 | 9 | 6 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 6 | 25
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 3 | 16
  Male | 3 | 3 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 6
  Not Hispanic or Latino | 8 | 7 | 4 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 8 | 4 | 20
  White | 1 | 1 | 2 | 4
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Participant With Treatment Emergent Adverse Events (TEAEs)
Description: Treatment-emergent adverse event, which is an undesirable event that occurs during or shortly after treatment begins.
Time Frame: Up to day 71
Measure: Count of Participants; unit: Participants
Groups:
- 2 mg/kg XTMAB-16: Single IV Infusion of 2 mg/kg XTMAB-16
- 4 mg/kg XTMAB-16: Single IV Infusion of 4 mg/kg XTMAB-16
- Pooled Placebo: Single IV Infusion of Placebo
Arm/Group | 2 mg/kg XTMAB-16 | 4 mg/kg XTMAB-16 | Pooled Placebo
Number analyzed (Participants) | 10 | 9 | 6
Participants | 2 | 3 | 1

2. Secondary Outcome: Participants by Cohort Who Test Positive for XTMAB-16 Anti-drug Antibody (ADA)
Description: Participants by cohort who test positive for XTMAB-16 ADA
Time Frame: ADA and nAB: Days 1, 8, 15, 29, 43, 57, 71
Measure: Count of Participants; unit: Participants
Arm/Group | 2 mg/kg XTMAB-16 | 4 mg/kg XTMAB-16 | Pooled Placebo
Number analyzed (Participants) | 10 | 9 | 6
Participants
  Day 1 ADA Screening | 0 | 0 | 0
  Day 8 ADA Screening | 0 | 0 | 0
  Day 15 ADA Screening | 1 | 1 | 0
  Day 15 ADA Confirmatory | 0 | 0 | 0
  Day 29 ADA Screening | 1 | 0 | 0
  Day 29 ADA Confirmatory | 1 | 0 | 0
  Day 43 ADA Screening | 4 | 0 | 0
  Day 43 ADA Confirmatory | 3 | 0 | 0
  Day 57 ADA Screening | 6 | 1 | 0
  Day 57 ADA Confirmatory | 5 | 1 | 0
  Day 71 ADA Screening | 6 | 3 | 0
  Day 71 ADA Confirmatory | 6 | 2 | 0

3. Secondary Outcome: Participants by Cohort Who Test Positive for XTMAB-16 Neutralizing Antibody (nAb)
Description: Participants by cohort who test positive for XTMAB-16 nAb
Time Frame: ADA and nAB: Days 1, 8, 15, 29, 43, 57, 71
Measure: Count of Participants; unit: Participants
Arm/Group | 2 mg/kg XTMAB-16 | 4 mg/kg XTMAB-16 | Pooled Placebo
Number analyzed (Participants) | 10 | 9 | 6
Participants
  Day 29 | 1 | 0 | 0
  Day 43 | 3 | 0 | 0
  Day 57 | 5 | 1 | 0
  Day 71 | 6 | 2 | 0

4. Secondary Outcome: XTMAB-16 Maximum Observed Concentration (Cmax)
Description: XTMAB-16 (Cmax)
Time Frame: Up to day 71
Measure: Mean (Standard Deviation); unit: Cmax (μg/mL)
Arm/Group | 2 mg/kg XTMAB-16 | 4 mg/kg XTMAB-16
Number analyzed (Participants) | 10 | 9
Cmax (μg/mL) | 64.17 (9.94) | 131 (23.42)

5. Secondary Outcome: XTMAB-16 Serum Observed Plasma Concentration at the End of Infusion (CT) Day 1
Description: XTMAB-16 serum (CT) Day 1
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: CT (μg/mL)
Arm/Group | 2 mg/kg XTMAB-16 | 4 mg/kg XTMAB-16
Number analyzed (Participants) | 10 | 9
CT (μg/mL) | 62.18 (6.757) | 128.9 (22.39)

6. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) XTMAB-16
Description: Time to maximum observed concentration (tmax) XTMAB-16
Time Frame: PK: Days 1, 2, 3, 4, 8, 15, 29, 43, 57, 71
Measure: Median (Full Range); unit: tmax (h)
Arm/Group | 2 mg/kg XTMAB-16 | 4 mg/kg XTMAB-16
Number analyzed (Participants) | 10 | 9
tmax (h) | 2.16 [2.1 to 8.65] | 3.0 [2.12 to 8.02]

7. Secondary Outcome: Area Under the XTMAB-16 Concentration-time Curve From Time Zero (Predose) Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-∞)
Description: Area under the XTMAB-16 concentration-time curve from time zero (predose) AUC0-∞
Time Frame: PK: Days 1, 2, 3, 4, 8, 15, 29, 43, 57, 71
Measure: Mean (Standard Deviation); unit: AUC0-inf (day*μg/mL)
Arm/Group | 2 mg/kg XTMAB-16 | 4 mg/kg XTMAB-16
Number analyzed (Participants) | 8 | 9
AUC0-inf (day*μg/mL) | 601.5 (231.8) | 1249 (245.0)

8. Secondary Outcome: Area Under the XTMAB-16 Concentration-time-curve From Time Zero to (Predose) Area Under the Plasma Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUC0-t)
Description: Area under the XTMAB-16 concentration-time-curve from time zero to (predose) AUC0-t
Time Frame: PK: Days 1, 2, 3, 4, 8, 15, 29, 43, 57, 71
Measure: Mean (Standard Deviation); unit: AUC0-last (day*μg/mL)
Arm/Group | 2 mg/kg XTMAB-16 | 4 mg/kg XTMAB-16
Number analyzed (Participants) | 9 | 9
AUC0-last (day*μg/mL) | 525.2 (238.0) | 1224 (235.9)

9. Secondary Outcome: Systemic Clearance After IV Dosing (CL)
Description: Systemic clearance after IV dosing (CL)
Time Frame: Up to day 71
Measure: Mean (Standard Deviation); unit: CL (L/day)
Arm/Group | 2 mg/kg XTMAB-16 | 4 mg/kg XTMAB-16
Number analyzed (Participants) | 8 | 9
CL (L/day) | 0.2498 (0.04883) | 0.2449 (0.06064)

10. Secondary Outcome: Apparent Terminal Half-life (t1/2)
Time Frame: Up to day 71
Measure: Mean (Standard Deviation); unit: t1/2 (day)
Arm/Group | 2 mg/kg XTMAB-16 | 4 mg/kg XTMAB-16
Number analyzed (Participants) | 8 | 9
t1/2 (day) | 8.644 (4.726) | 10.23 (3.617)

11. Secondary Outcome: Volume of Distribution Following IV Dosing (Vz) Day 1 up to Day 71
Time Frame: Up to day 71
Measure: Mean (Standard Deviation); unit: Vz (L)
Arm/Group | 2 mg/kg XTMAB-16 | 4 mg/kg XTMAB-16
Number analyzed (Participants) | 8 | 9
Vz (L) | 2.864 (0.8861) | 3.435 (0.9878)

12. Secondary Outcome: Mean Residence Time (MRT)
Description: Mean residence time (MRT)
Time Frame: Up to day 71
Measure: Mean (Standard Deviation); unit: MRT (day)
Arm/Group | 2 mg/kg XTMAB-16 | 4 mg/kg XTMAB-16
Number analyzed (Participants) | 8 | 9
MRT (day) | 12.51 (6.214) | 13.32 (3.794)

ADVERSE EVENTS:
Time Frame: The Investigator or designee recorded all reportable events with start dates occurring from informed consent until 7 (for nonserious AEs) or 30 days (for SAEs) after the last day of study participation. Study participation was up to 71 days.
Arm/Group | 2 mg/kg XTMAB-16 | 4 mg/kg XTMAB-16 | Pooled Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/9 | 0/6
Other Adverse Events (participants affected / at risk) | 3/10 | 4/9 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 mg/kg XTMAB-16 (N=10) | 4 mg/kg XTMAB-16 (N=9) | Pooled Placebo (N=6)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 mg/kg XTMAB-16 (N=10) | 4 mg/kg XTMAB-16 (N=9) | Pooled Placebo (N=6)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Emesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter Site Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Eye Pain due to Covid Testing (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lightheadedness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Loose Stool (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Foggy Feeling (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/95/NCT04971395/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/95/NCT04971395/SAP_001.pdf